CLINICAL TRIAL: NCT02390700
Title: Golimumab Intravenous Infusion Registry (GO-IV)
Brief Title: Observational Study of Golimumab Intravenous Infusion
Acronym: GO-IV
Status: Terminated | Type: Observational
Why Stopped: Business decision based on lack of enrollment
Sponsor: Janssen Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: CR105631; CNTO148ARA4003 (Other: Janssen Inc.)
Record Dates: First submitted 2015-03-11; First posted 2015-03-17 (Estimated); Last update posted 2016-11-17 (Estimated); Status verified 2016-11

CONDITIONS: Rheumatoid Arthritis
Keywords: Rheumatoid Arthritis; Observational; Golimumab; SIMPONI; Intravenous Infusion
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — golimumab

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Golimumab Intravenous: Participants with rheumatoid arthritis (RA) in Canada, will be observed for 24 months. Only data available from source documentation will be collected.
  Interventions: Biological: Golimumab Intravenous

INTERVENTIONS:
Biological: Golimumab Intravenous — This is a non-interventional study. Participants with rheumatoid arthritis in Canada will be observed for 24 months.
  Other Names: SIMPONI

SUMMARY:
The purpose of this study is to evaluate the incidence and management of infusion reactions with Golimumab intravenous infusion.

DETAILED DESCRIPTION:
This is a prospective, observational, non-interventional (no treatment given during course of the study) multi-center (when more than one hospital or medical school team work on a medical research study), study that will enroll participants with rheumatoid arthritis (RA) in Canada. Only data available from source documentation will be collected. The participation in this study will not impact on the standard of care of the participant or any benefits to which they are otherwise entitled. All aspects of treatment decisions and clinical management of participants will be in accordance with clinical practice and at the discretion of the health care provider. Participants' safety will be monitored throughout the study.

ELIGIBILITY:
Inclusion Criteria:

* Participants must have a confirmed diagnosis of rheumatoid arthritis
* Participants must have provided a written consent for data collection by signing an informed consent form indicating that he/she understand the purpose and procedures for data collection and are willing to participate in the study
* Participants are golimumab-naive (never have used golimumab both SC and IV formulations)
* Participants are prescribed golimumab intravenous by an appropriate physician as per the Canadian Product Monograph

Exclusion criteria:

* Participant who has been treated with golimumab in the past
* Participant has been diagnosed with psoriatic arthritis or ankylosing spondylitis
* Participant has received an investigational drug (including investigational vaccines) or used an invasive investigational medical device within 30 days before the start of the study or first data collection time point
* Participant is currently enrolled in an interventional study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Canadian participants with rheumatoid arthritis (RA), who have been prescribed intravenous golimumab prior to, and independently of, study enrollment.
Sampling Method: Non-Probability Sample
Enrollment: 78 (Actual)
Dates: Start 2015-02; Primary Completion 2016-10 (Actual); Study Completion 2016-10 (Actual)

PRIMARY OUTCOMES:
Number of Participants With Infusion Reactions | Up to end of study (2 years) or early withdrawal
  The count of infusion reactions will be reported.

SECONDARY OUTCOMES:
Number of Participants With use of Pre-infusion Medications | Baseline up to end of study (2 years) or early withdrawal
  Participants with administration of Pre-infusion medications or combination of Pre-infusion medications will be reported. The list of pre-treatments includes: acetaminophen, anti-histamines, steroids (Hydrocortisone, Prednisone), acetaminophen alone, anti-histamines alone, steroids alone, steroids + anti-histamines, steroids + acetaminophen, anti-histamines + acetaminophen, steroids + anti-histamines + acetaminophen.
Number of Participants With use of Concomitant Medications at Time of Infusion | Baseline up to end of study (2 years) or early withdrawal
  Participants with type of concomitant medications used at time of infusion will be reported. The groups of concomitant medication of interest are: any immunosuppressant (IS), methotrexate and corticosteroids.
Number of Participants With Infusion Reaction Treatments | Baseline up to end of study (2 years) or early withdrawal
  For each infusion administration with infusion reactions, type of medications was used to treat the reaction will be reported. The list of medications includes anti-histamines, steroids, and epinephrine.
Number of Participants With Subsequent Reactions After the First Infusion Reaction | Baseline up to end of study (2 years) or early withdrawal
  For each participant who has experienced at least 1 infusion reaction after enrolment, occurrence of infusion reaction at subsequent infusions after the first infusion reaction will be assessed.
Change From Baseline in Rheumatoid Arthritis Impact of Disease (RAID) Score | Baseline up to end of study (2 years) or early withdrawal
  The RAID is self-administered questionnaire which includes seven domains (pain, function, fatigue, physical and psychological wellbeing, sleep disturbance and coping). Each domain is evaluated using a single question answered by a 0 to 10 numerical rating scale. Each domain also has a specific weight assigned by a patient survey. The RAID score is a continuous variable ranging from 0 (best) to 10 (worst).
Percentage of Participants With Absolute Change of at Least 3 Points in RAID Score | Baseline up to end of study (2 years) or early withdrawal
  The RAID is self-administered questionnaire which includes seven domains (pain, function, fatigue, physical and psychological wellbeing, sleep disturbance and coping). Each domain is evaluated using a single question answered by a 0 to 10 numerical rating scale. Each domain also has a specific weight assigned by a patient survey. The RAID score is a continuous variable ranging from 0 (best) to 10 (worst).
Percentage of Participants With Relative Change of at Least 50 Percent (%) and a Maximum Score of 2 in RAID Score | Baseline up to end of study (2 years) or early withdrawal
  The RAID is self-administered questionnaire which includes seven domains (pain, function, fatigue, physical and psychological wellbeing, sleep disturbance and coping). Each domain is evaluated using a single question answered by a 0 to 10 numerical rating scale. Each domain also has a specific weight assigned by a patient survey. The RAID score is a continuous variable ranging from 0 (best) to 10 (worst).

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Inc. Clinical Trial, Study Director — Janssen Inc.
Locations (13):
- Canada (13):
  - St. John's, Newfoundland and Labrador
  - Ancaster, Ontario
  - Barrie, Ontario
  - Kitchener, Ontario
  - Mississauga, Ontario
  - Nepean, Ontario
  - Oakville, Ontario
  - St. Catharines, Ontario
  - Toronto, Ontario
  - Laval, Quebec
  - Montreal, Quebec
  - Saskatoon, Saskatchewan
  - Victoria